CLINICAL TRIAL: NCT02114281
Title: Oral and Dental Health Status in Patients Suffering From Chronic Kidney Disease
Acronym: NEPHRODENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2013/11
Record Dates: First submitted 2014-02-04; First posted 2014-04-15 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Chronic Kidney Disease
Keywords: Oral Health; Periodontitis; Tooth cavities; Saliva; Halitosis; Mucosa; Chronic kidney disease; Inflammation; Nutrition
MeSH Terms: conditions — Renal Insufficiency, Chronic; Periodontitis; Dental Caries; Halitosis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care (Experimental): Patient with dental care
  Interventions: Other: Care
- Not care (Active Comparator): Patient with not dental care
  Interventions: Other: Not care

INTERVENTIONS:
Other: Care
  Arms: Care
Other: Not care
  Arms: Not care

SUMMARY:
A large panel of oral and dental diseases exist in patients suffering from chronic kidney disease (CKD) in end-stage renal disease: it concerns teeth, peridontium, alveolar bone and saliva and it has been already described in the literature. The consequences of oral diseases in systemic health are substantial, including increase of inflammatory parameters, alteration of nutrition and increase of cardiovascular risk factors. It has been shown before that several oral diseases can be considered as cardiovascular risk factor in the general population and in diabetic patients through the chronic inflammatory pathway. In CKD patients, the influence of oral diseases on the progression of the chronic kidney disease is not yet established, as most of the studies are focused on stage 5 CKD or dialysis patients. That's why the interactions between dental health and CKD will be evaluated in this population of patients, at different stages of the disease (stages 2 to 5).

The main objective will be to describe the oral diseases at each stage of CKD. Secondary objectives will be: (1) To evaluate the link between the oral health and the chronic kidney disease stage, the nutritional and inflammatory status; (2) Among patients needing dental treatments, to evaluate after 6 months and 12 months whether dental cares have an influence on nutrition parameters, inflammatory status and CKD; (3) to evaluate the completion of dental treatments after the dental consultation including advises on dental health.

DETAILED DESCRIPTION:
The consequences of oral and dental diseases in general health are substantial, including acute infectious process starting from teeth or peridontium, benign or malignant diseases starting from mucosa or teeth/peridontium and an overall reduction of nutrition indices and a decrease of quality of life markers. More recently, an augmentation of systemic inflammatory reaction markers has been shown correlated with periodontal diseases, leading to an increase of cardiovascular diseases and/or diabetic risk in those patients. A large panel of oral and dental diseases has been described in patients suffering from chronic kidney disease (CKD) in a terminal stage or dialysis (haemodialysis and peritoneal dialysis). In CKD patients, the influence of oral diseases on the progression of the chronic kidney disease is not established today, as most of the studies are focused on stage 5 CKD or dialysis patients. That's why the interactions between dental health and CKD will be evaluated in these patients, at different stages of the disease (stages 2 to 5). In this study, it is hypothesized that the augmentation of inflammation and the alteration of nutrition due to oral diseases have an impact on the alteration of CKD patients, through the chronic inflammatory pathway. We will evaluate the oral and dental health at Day 0, 6 months and 12 months using several indices: the oral hygiene-simplified index, the community periodontal index in treatment needs index, the decayed missing filled per tooth index, the number of functional teeth index, the oral health impact profile index, the saliva composition, the evaluation of halitosis and a mucosa evaluation. In parallel, an evaluation of the influence of chronic oral diseases on nutrition, inflammation and progression of chronic kidney disease will be done: biological check-up, nutrition intake statement and body mass index.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients, stage 2 to 5, under treatment in CHU de Bordeaux
* Aged more than 18 years old
* A free, informed and written consent will be established
* Must have a medical plan
* Patients have had no dental cares 6 months before the inclusion date

Exclusion Criteria:

* Persons having a current law affair
* Persons suffering from psychosis or severe mental impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Evolution of the status of oral health, which will be evaluated through several dental epidemiological indices (composite measure) | 12 months after the inclusion
  The primary outcome is a composite measure including :
  * Oral Hygiene Index-Simplified index (OHI-S)
  * Community Periodontal Index in Treatment Needs index (CPITN)
  * Decayed Missing Filled per Tooth Index (DMF-T)
  * Number of Functional Teeth index (FS-T)
  * Oral Health Impact Profile index (OHIP)
  * Saliva Check (stimulated and non stimulated saliva flow, pH, buffer activity)
  * Halitosis evaluation (quantification of sulfur volatils compounds)
  * Mucosa evaluation

SECONDARY OUTCOMES:
Evolution of nutrition statement | 12 months after the inclusion
  food survey, biological assessment and body composition by bioelectrical impedance analysis
Evolution of chronic inflammation | 12 months after the inclusion
Progression of chronic kidney disease (CKD) | 12 months after the inclusion
Compliance with dental treatments in CKD patients | 12 months after the inclusion
Evolution of CKD diseases with/without dental treatments in those patients who need dental treatments | 12 months after the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Claire RIGOTHIER, MD, Principal Investigator — University Hospital Bordeaux, France; Antoine BENARD, MD, Study Chair — University Hospital Bordeaux, France
Locations (1):
- Service de néphrologie, transplantation et dialyse - Hôpital Pellegrin, Bordeaux, France